CLINICAL TRIAL: NCT01779388
Title: Role of Bronchoscopy Assisted by Electromagnetic Navigation (EMN) in the Diagnosis of Small Pulmonary Nodules of Indeterminate Nature. A Prospective Study by the European Lung Cancer Working Party.
Brief Title: Bronchoscopy Assisted by Electromagnetic Navigation (EMN) in the Diagnosis of Small Pulmonary Nodules
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European Lung Cancer Working Party (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 01201
Record Dates: First submitted 2013-01-28; First posted 2013-01-30 (Estimated); Last update posted 2022-04-04 (Actual); Status verified 2021-08

CONDITIONS: Pulmonary Nodule Cm
Keywords: Lung nodule; PET scanner; Bronchoscopy; Electromagnetic navigation
MeSH Terms: interventions — Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bronchoscopy guided by fluoroscopy (Other): Bronchoscopy guided by fluoroscopy followed by ENG
  Interventions: Procedure: Bronchoscopy
- Bronchoscopy guided by electromagnetic navigation (Experimental): Bronchoscopy guided by ENG followed by fluoroscopy
  Interventions: Procedure: Bronchoscopy

INTERVENTIONS:
Procedure: Bronchoscopy — During a general anaesthesia, an evaluation will be done by conventional bronchoscopy guided by fluoroscopy and by bronchial endoscopy guided by electromagnetic navigation, the selection of order in techniques being randomly assigned.

SUMMARY:
Due to CT screening, a lot of peripheral nodule not accessible to conventional endoscopy will be found. Electromagnetic navigation directed bronchoscopy (ENB) is a new technique needing validation. the primary aim of the study is to compare ENB to radiologically guided bronchoscopy, considered the standard comparator.

ELIGIBILITY:
Inclusion Criteria:

* Presence on a conventional or low dose chest CT at least one lung nodule 5-20 mm in its largest axis, of indeterminate nature; the nodule must be positive at PET-CT examination (in case of PET-CT negative, only follow-up is proposed)
* The pulmonary nodule(s) must be known for less than 6 months
* The nodule appearance can be solid, presents as a ground glass opacity with solid component or as pure ground glass opacity
* Availability for participating in the detailed follow-up of the protocol
* Signed informed consent.
* Age > 18 years

Exclusion Criteria:

* Nodules found in the context of an active infection or for whom, the clinical context and/or additional available investigations (serology, microbiological samplings, immune abnormalities) show that cancer diagnosis is unlikely
* Nodules found in the context of an active previously documented disease that can be associated with pulmonary nodules (anthracosilicosis, histoplasmosis, tuberculosis, autoimmune or rheumatoid diseases …)
* Calcified nodule
* Anticoagulation therapy of any type that cannot be suspended for the duration of the investigation
* Respiratory failure, recent myocardial infarction (less than 3 months prior to the date of lung nodule screening), uncontrolled angina pectoris, congestive cardiac failure, cardiac arrhythmia, uncontrolled infectious disease or any other physical, biological or psychological factor which may prevent adherence to the study protocol or which may impair the patient's tolerance to the endoscopy and/or the general anaesthesia
* Presence of a implanted cardiac device (pace-maker, defibrillator, …)
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-01 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Capability of diagnosing lung nodule with ENB (Sensitivity) | After the procedure
  Calculate the sensitivity of each endoscopic technique in obtaining the diagnostic of the pulmonary nodule

SECONDARY OUTCOMES:
Prediction of malignancy | After the procedure
  To identify a predictive molecular signature able to predict the malignant nature of the nodule by studying the transcriptome (miRNAs and mRNAs) and the single nucleotide polymorphism (SNPs) by using high throughput techniques in biopsies, alveolar lavage, blood and exhaled breath

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Berghmans, MD, PhD, Study Chair — ELCWP; Dimitri Leduc, MD, PhD, Principal Investigator — ELCWP
Locations (1):
- Institut Jules Bordet, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided